CLINICAL TRIAL: NCT02867930
Title: Comparative Effects of Dexmedetomidine and Ketofol for Sedation in Out-patients Undergoing Diagnostic Trans-esophageal Echocardiography: A Randomized Controlled Trial
Brief Title: Comparative Effects of Dexmedetomidine and Ketofol for Sedation in Patients Undergoing Trans-esophageal Echocardiography
Acronym: KDTEE
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Post Graduate Institute of Medical Education and Research, Chandigarh (Other)
Responsible Party: Principal Investigator, Sruthi Sankar, Post graduate student Junior resident, Post Graduate Institute of Medical Education and Research, Chandigarh
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: KDTEE16
Record Dates: First submitted 2016-06-30; First posted 2016-08-16 (Estimated); Last update posted 2017-11-06 (Actual); Status verified 2017-11

CONDITIONS: Heart Valve Disease; Heart Septal Defects, Atrial
Keywords: Echocardiography; Transesophageal; Dexmedetomidine; Ketamine; Propofol
MeSH Terms: conditions — Heart Valve Diseases; Heart Septal Defects, Atrial | interventions — Dexmedetomidine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group D (Active Comparator): Dexmedetomidine- drug used for moderate sedation prepared as 200 mic in 20 ml syringe.with intravenous loading dose at 1ml/kg/hour till required sedation is achieved and maintenance infusion of 0.05mg/kg/hour till completion of transesophageal echocardiography
  Interventions: Drug: Dexmedetomidine
- Group KF (Active Comparator): Ketamine+Propofol -drugs used for sedation-as ratio 1:3with 19ml of 1% propofol + 1.3ml ketamine(50mg/ml) as loading intravenous infusion dose at 1ml/kg/hour till required sedation is achieved and maintenance infusion of 0.05mg/kg/hour till completion of transesophageal echocardiography
  Interventions: Drug: Ketofol(ketamine+propofol)

INTERVENTIONS:
Drug: Dexmedetomidine — drug for moderate sedation in trans-esophageal echocardiography
  Arms: Group D
Drug: Ketofol(ketamine+propofol) — drug for moderate sedation in trans-esophageal echocardiography
  Arms: Group KF

SUMMARY:
The purpose of the study is to compare dexmedetomidine and ketofol to find a suitable alternative for moderate sedation in out-patient diagnostic trans-esophageal echocardiography.

DETAILED DESCRIPTION:
Sample size was estimated based on previous studies with sedation in equally invasive procedures that in 2 groups difference in time to achieve Ramsay sedation scale was 0.8min.(In group dexmedetomidine 12.4 & group ketofol 13.2 with S.D of 0.8). The sample size came out to be 22 subjects per group at a power of 90 % & confidence interval of 95 %. For possible dropouts, it was decided to include 10% extra subjects so finally it was decided to include 25 subjects per group. (Total sample size 50 subjects)

Normality of quantitative data will be checked by measures of Kolmogorov Smirnov tests of normality. If data is normally distributed Student t-test will be applied for comparison of 2 groups. Mann-Whitney U-test will be used for statistical analysis of skewed continuous variables or ordered categorical data. Proportions will be compared using Chi square or Fisher's exact test whichever is applicable. Wilcoxon Signed rank test will be used for skewed data or for scores (time related variables). . For comparison (time related variables) of Hemodynamics Repeated Measure ANOVA will be applied. All statistical tests will be two-sided and will be performed at a significance level of α=0.05. Analysis will be conducted using SPSS for Windows

ELIGIBILITY:
Inclusion Criteria:

* Patients with Atrial septal defect/Valvular Heart disease (MS/MR/AS/AR)

Exclusion Criteria:

* Atrial fibrillation with fast ventricular rate
* Congestive cardiac failure
* BMI > 30
* Perforated viscus/active GI bleed
* Esophageal stricture/tumor/laceration
* H/o radiation to neck & mediastinum
* H/o GI surgery or H/o dysphagia
* Restriction of neck mobility
* Active esophagitis/peptic ulcer disease
* Symptomatic bradycardia
* Seizure disorder
* Coagulopathy/thrombocytopenia

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2016-06; Primary Completion 2016-12 (Actual); Study Completion 2016-12-30 (Actual)

PRIMARY OUTCOMES:
Time taken to achieve adequacy of sedation before probe insertion. | maximum of 10 minutes
  Adequacy of sedation to be measured using Ramsay Sedation Scale (>=3 considered adequate for probe insertion)

SECONDARY OUTCOMES:
Recovery time | Upto 30 minutes
  Time to achieve modified aldrete score >9
Heart rate during procedure | every 5 minutes till end of procedure
  Heart rate in beats/min, , facial pain score as 0-10
mean arterial pressure during procedure | every 5 minutes till end of procedure
  mean arterial pressure in mmHg,
Oxygen saturation during procedure | every 5 minutes till end of procedure
  oxygen saturation in %
End tidal carbondioxide during procedure | every 5 minutes till end of procedure
  End tidal carbon dioxide in mm Hg

CONTACTS AND LOCATIONS:
Overall Officials: Sruthi Sankar, Principal Investigator — Post Graduate Institute of Medical Education and Research, Chandigarh
Locations (1):
- Postgraduate Institute of Medical Education and Research, Chandigarh, India

IPD SHARING:
Plan to Share IPD: Undecided